CLINICAL TRIAL: NCT06078709
Title: Preoperative Hypofractionated Radiotherapy With FOLFOX for Esophageal/Gastroesophageal Junction Adenocarcinoma (PHOX)
Brief Title: Preoperative Hypofractionated Radiotherapy With FOLFOX for Esophageal or Gastroesophageal Junction Adenocarcinoma
Acronym: PHOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2241; NCI-2023-07432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GMROR2241 (Other: Mayo Clinic Radiation Oncology); 23-001689 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage I Esophageal Adenocarcinoma AJCC v8; Clinical Stage I Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: interventions — Specimen Handling; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Endoscopy, Digestive System; Gastroscopy; Fluorouracil; dehydroftorafur; Radiation Dose Hypofractionation; Radiation; Leucovorin; Oxaliplatin; Magnetic Resonance Spectroscopy; X-Rays; Docetaxel; durvalumab; Disulfides; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (FLOT and Radiation and FOLFOX) (Experimental): Patients received Induction Chemotherapy [FLOT (5-FU/leucovorin/oxaliplatin/docetaxel)] following by radiation therapy daily for 3 weeks with 2 concurrent cycles of FOLFOX per protocol. See detailed description for more information.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Endoscopic Ultrasound; Procedure: Esophagogastroduodenoscopy; Drug: Fluorouracil; Radiation: Hypofractionated Radiation Therapy; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Other: Survey Administration; Drug: Docetaxel; Biological: Durvalumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT and PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography; Computerized Tomography (CT) scan
Procedure: Endoscopic Ultrasound — Undergo EUS
  Other Names: endosonography; EUS
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD; Upper Endoscopy
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757; 2,4-Dioxo-5-fluoropyrimidine; 51-21-8
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669; JM83; RP54780; SR96669
Procedure: Positron Emission Tomography — Undergo PET and PET/CT scan
  Other Names: Medical Imaging; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Survey Administration — Ancillary studies
Drug: Docetaxel — Given IV
  Other Names: 148408-66-6; Docecad; N-Debenzoyl-N-(tert-butoxycarbonyl)-10-deacetyltaxol; RP 56976; RP-56976; RP56976; Taxotere
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; MEDI 4736; MEDI-4736; MEDI4736; Disulfide with Human Monoclonal MEDI4736 Kappa-chain; Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain); Immunoglobulin G1

SUMMARY:
This phase II trial tests how well preoperative (prior to surgery) radiation therapy with fluorouracil, oxaliplatin, and leucovorin calcium (FOLFOX) works for the treatment of stage I-III esophageal or gastroesophageal junction adenocarcinoma. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Fluorouracil stops cells from making deoxyribonucleic acid (DNA) and it may kill tumor cells. Leucovorin is not a chemotherapy medication but is given in conjunction with chemotherapy. Leucovorin is used with the chemotherapy medication fluorouracil to enhance the effects of the fluorouracil, in other words, to make the drug work better. Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It damages the cell's DNA and may kill tumor cells. Giving preoperative hypofractionated radiation with fluorouracil and oxaliplatin may kill more tumor cells in patients with stage I-III esophageal or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate non-inferiority of pathologic complete response (pCR) with hypofractionated radiotherapy and concurrent FOLFOX compared to historical controls.

SECONDARY OBJECTIVES:

I. Report targeted acute grade ≥ 3 gastrointestinal (GI) toxicity, per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

II. Assess post-operative toxicity for patients undergoing esophagectomy, as determined by the Clavien-Dindo Classification.

III. Analyze patient-reported quality of life, per Functional Assessment of Cancer Therapy- Esophageal (FACT-E).

IV. Determine the financial toxicity of hypofractionated radiotherapy, using Comprehensive Score for Financial Toxicity (COST-FACIT).

V. Report overall survival and progression-free survival. VI. Report long-term toxicity secondary to trimodality therapy. VII. Report event-free survival. VIII. Assess outcomes for patients treated with hypofractionated radiotherapy and FOLFOX but who did not proceed to esophagectomy.

IX. Compare toxicity of chemoradiation between patients receiving proton based versus (vs.) photon-based radiotherapy.

X. Compare clinical outcomes and pCR for patients receiving hypofractioned radiotherapy but different induction chemo (immuno) therapy regimens: no induction vs. fluorouracil, oxaliplatin, leucovorin, docetaxel (FLOT) vs. FLOT + durvalumab.

CORRELATIVE OBJECTIVES:

I. Explore the predictive and prognostic role for circulating tumor DNA in esophageal cancer.

II. Study the utility of whole exome and germline sequencing to predict chemoradiation treatment response.

III. Explore the predictive power of whole exome sequencing regarding chemoradiotherapy toxicity.

IV. Implement whole exome and germline sequencing to personalize immunotherapy in esophageal cancer.

V. Study the predictive and prognostic role of tumor-derived extracellular vesicles in esophageal cancer.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive 5-FU intravenously (IV) over 24 hours on day 1, leucovorin calcium IV over 10-120 minutes on day 1, oxaliplatin IV over 2-6 hours on day 1, and docetaxel IV over 1 hour on day 1 of each cycle. Treatment repeats every 2 weeks for a total of up to 6 cycles in the absence of disease progression or unacceptable toxicity. Eligible patients also receive durvalumab IV over 1 hour every 4 weeks in the absence of disease progression or unacceptable toxicity. After completion of FLOT, patients undergo radiation therapy daily for 3 weeks with 2 concurrent cycles of FOLFOX.

FOLFOX: Patients receive oxaliplatin IV over 2-6 hours on day 1, leucovorin calcium IV over 10-120 minutes on day 1, and and fluorouracil IV over 46-48 hours on days 1 and 2. of each cycle. Treatment repeats every 2 weeks for a total of 3 cycles in the absence of disease progression or unacceptable toxicity. Starting at cycle 2, patients undergo radiation therapy daily on Monday through Friday for a total of 15 treatments. Patients undergo esophagogastroduodenoscopy (EGD) and/or endoscopic ultrasound (EUS) during screening and undergo computed tomography (CT)/position emission tomography (PET) scan and CT scan as well as blood and tissue sample collection throughout the study.

After completion of study treatment, patients are followed up at 6,12 and 24 months and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of esophageal or gastroesophageal junction adenocarcinoma, American Joint Committee on Cancer (AJCC) 8th edition stage T1-4N0-3M0
* Candidate for trimodality therapy: neoadjuvant chemo (immuno) therapy, chemoradiation, and esophagectomy
* Surgical consultation has confirmed that patient is an appropriate candidate for esophagectomy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Negative pregnancy test done ≤ 7 days prior to chemotherapy, for women of childbearing potential only
* Ability to provide written informed consent and complete questionnaire(s) by themselves or with assistance
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood and tissue samples for correlative research purposes

Exclusion Criteria:

* Clinical or biopsy-proven distant metastatic disease (AJCC 8th edition stage TanyNanyM1)
* Cervical or upper esophageal tumor
* Prior chemotherapy or radiotherapy for esophageal cancer or history of radiotherapy to the thorax
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgement of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with proper assessment of adverse events
* Receiving any investigational agent which would be considered as a treatment for the primary neoplasm or other active malignancy ≤ 1 year prior to registration that is considered by the investigator to interfere with the current treatment or measurement of outcomes
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Up to 5 years after completion of chemoradiation
  A single-group design will be used to test whether the proportion is potentially non-inferior, with a non-inferiority proportion (P0) of 0.13 (H0: P ≤ 0.13 versus H1: P > 0.13).

SECONDARY OUTCOMES:
Incidence of acute ≥ gastrointestinal (GI) adverse events (AEs) | Up to 6 weeks after completion of chemoradiation
  Report acute grade ≥ 3 GI AEs per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. Will be summarized descriptively.
Incidence of post operative AEs | From surgery up to 6 months after completion of chemoradiation
  Determined by the Clavien-Dindo Classification. Will be summarized descriptively.
Patient-reported quality of life (QOL) | Up to 24 months after completion of chemoradiation
  Per Functional Assessment of Cancer Therapy- Esophageal. Will be assessed over time. Wilcoxon signed-rank tests will be used to calculate p-values. Descriptive statistics and graphical methods will also be used to summarize the data.
Financial toxicity | Up to 24 months after completion of chemoradiation
  Financial toxicity will be measured using the COmprehensive Score for financial Toxicity (COST), a patient-reported outcome measure that describes the financial distress experienced by cancer patients. The survey consists of 12 questions, each answered with a 0-4 scale where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, and 4=Very much. Results will be reported descriptively and include separate consideration of individual item scores.
Overall survival (OS) | From study entry to death from any cause, up to 5 years after completion of chemoradiation
  Will be assessed graphically using the Kaplan-Meier method. Summary statistics will be reported, including medians, 95% confidence intervals, etc.
Progression-free survival (PFS) | From study entry to the first of either disease progression or death, up to 5 years after completion chemoradiation
  Will be assessed graphically using the Kaplan-Meier method. Summary statistics will be reported, including medians, 95% confidence intervals, etc.
Long-term toxicity secondary to trimodality therapy | Up to 5 years after completion of chemoradiation
  Will be reported descriptively using CTCAE version 5.0 criteria.
Event free survival | From study entry to the first of either disease progression or recurrence or relapse or death, up to 5 years after completion of chemoradiation
  Will be assessed graphically using the Kaplan-Meier method. Summary statistics will be reported, including medians, 95% confidence intervals, etc.
Outcomes for patients treated with hypofractionated radiotherapy and FOLFOX but who did not proceed to esophagectomy | Up to 5 years after completion of chemoradiation
  OS and PFS will be assess using Kaplan-Meier methodology. Summary statistics will be reported, including medians, 95% confidence intervals, etc. AEs and QOL data will be reported with summary statistics and graphical methods, as appropriate.
Toxicity of chemoradiation between patients receiving proton based versus photon-based radiotherapy | Up to 5 years after completion of chemoradiation
  Will be done descriptively, reporting frequencies and percentages between patients.
Toxicity of chemoradiation between groups receiving proton based versus photon-based radiotherapy | Up to 5 years after completion of chemoradiation
  Will be done descriptively, reporting toxicity rates between groups using the chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L. Hallemeier, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials